CLINICAL TRIAL: NCT00857441
Title: A Prospective Three-arm Multi-center Study to Investigate Procedural, Clinical and Angiographic Outcomes Using a Drug Eluting Balloon Versus a Standard Balloon in Combination With a Bare Metal Stent and a DES Stent, Following the Provisional Side Branch T-stenting Approach, in Patients With Complex Lesions
Brief Title: Drug-eluting Balloon in Bifurcations Trial
Acronym: DEBIUT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Prof. Pieter Stella, Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRF8025
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Stable Angina; Unstable Angina
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Angina, Stable; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Use of Dior balloon and implant of Liberté Bare Metal Stent
  Interventions: Device: Drug eluting balloon; Device: Liberté
- 2 (Active Comparator): Use of standard balloon and implant of Liberté Bare Metal Stent
  Interventions: Device: Liberté; Device: PTCA balloon catheter
- 3 (Active Comparator): Use of standard balloon and implant of Taxus Liberté Drug Eluting Stent
  Interventions: Device: PTCA balloon catheter; Device: Taxus

INTERVENTIONS:
Device: Drug eluting balloon — Percutaneous transluminal coronary balloon angioplasty catheter eluting paclitaxel
  Other Names: Dior (EuroCor)
  Arms: 1
Device: Liberté — Bare metal stent
  Other Names: Liberté (Boston Scientific)
  Arms: 1; 2
Device: PTCA balloon catheter — Percutaneous transluminal coronary angioplasty catheter
  Other Names: Any PTCA catheter
  Arms: 2; 3
Device: Taxus — Paclitaxel eluting stent
  Other Names: Taxus Liberté (Boston scientific)
  Arms: 3

SUMMARY:
The purpose of the DEBIUT study is to assess procedural, clinical and angiographic outcomes of:

1. Provisional T-stenting use for dilation the Paclitaxel-eluting PCI-balloon (DiorTM) in comparison to dilation with a standard balloon prior to the implant of the Liberty Bare Metal Stent in bifurcation lesions (with side branch involvement).
2. Comparison of the results above with the results of using a standard balloon prior to provisional T-stenting with the Paclitaxel-eluting stent TaxusTM LibertéTM.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris (CCS class 1,2,3,4) or unstable angina and documented ischemia or silent ischemia
* Patients eligible for coronary revascularisation
* The target bifurcation lesion has a major native coronary artery (>2.5mm) with a stenosis > 50% (on visual assessment) located at a side branch (>2mm)
* Patient must be acceptable for CABG
* De novo lesion
* The main vessel lesion can be covered by one stent (up to 32mm)
* Only one target lesion can be included in the study: other lesions in different vessels are successfully treated before the treatment of the target lesion (residual stenosis <30%, stent well deployed, no residual dissection, normal TIMI flow, no chest pain, ECG unchanged compared to pre-procedural ECG)
* Signed patients informed consent

Exclusion Criteria:

* Patient unable to give informed consent
* Patients with a previous PCI in the target vessel
* Patients with in stent restenosis of target lesion
* Left ventricular ejection fraction more than 30%
* Patients with left main disease
* Severe calcifications with an undilatable lesion during balloon predilatation
* History of bleeding diathesis
* Untreated significant lesion greater than 50% diameter stenosis remaining proximal or distal to the target intervention.
* Patient has suffered a stroke or TIA within the past 3 months
* Life expectancy < 1 year
* Any major surgery planned or required during the next 6 months
* Acute Myocardial Infarction
* Only one target lesion can be included in the study
* Allergy to contrast and/or required anti-platelet medication
* Patients unwilling to return for follow-up at 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Side branch angiographic Late Lumen Loss (expressed in millimeters) measured by Quantitative Coronary Analysis (QCA) | 6 months

SECONDARY OUTCOMES:
Target vessel failure (TVF) | 6 months
Major Angiographic coronary or cerebral Events (MACCE) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Stella, MD, Principal Investigator — UMC Utrecht
Locations (3):
- Belgium (2):
  - Oost-Limburg Ziekenhuis, Genk
  - Gasthuisberg Leuven, Leuven
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Belkacemi A, Agostoni P, Voskuil M, Stella PR. Coronary bifurcation lesions treated with the drug-eluting balloon: a preliminary insight from the DEBIUT study. EuroIntervention. 2011 May;7 Suppl K:K66-9. doi: 10.4244/EIJV7SKA12. PMID 22027731